CLINICAL TRIAL: NCT00733993
Title: Experiment 1: Adenosine Receptor A2A Antagonists and Cocaine Dependence
Brief Title: Caffeine and Cocaine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Frederick Gerard Moeller, Professor - Division Chair, Addiction Psychiatry, Virginia Commonwealth University
Allocation: Non-Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: DA09262; P50DA009262 (NIH); DPMCDA
Record Dates: First submitted 2008-08-12; First posted 2008-08-13 (Estimated); Results first posted 2017-03-22 (Actual); Last update posted 2017-03-22 (Actual); Status verified 2017-02

CONDITIONS: Cocaine Dependence
Keywords: substance abuse; cocaine; caffeine; impulsivity
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders; Impulsive Behavior | interventions — Caffeine; Amphetamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 Caffeine 150 mg (Experimental): Caffeine 150 mg
  Interventions: Drug: Caffeine 150 MG
- 2 Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 3 Amphetamine (Experimental): Amphetamine
  Interventions: Drug: Amphetamine
- 4 Caffeine 300 mg (Experimental): Caffeine 300 mg
  Interventions: Drug: Caffeine 300 MG

INTERVENTIONS:
Drug: Caffeine 150 MG — Across five separate testing days, subjects were administered two placebo doses, 20 mg amphetamine, 150 mg caffeine, and 300 mg caffeine in counterbalanced fashion
  Other Names: Vivarin
  Arms: 1 Caffeine 150 mg
Drug: Placebo — Across five separate testing days, subjects were administered two placebo doses, 20 mg amphetamine, 150 mg caffeine, and 300 mg caffeine in counterbalanced fashion
  Arms: 2 Placebo
Drug: Amphetamine — Across five separate testing days, subjects were administered two placebo doses, 20 mg damphetamine,150 mg caffeine, and 300 mg caffeine in counterbalanced fashion
  Arms: 3 Amphetamine
Drug: Caffeine 300 MG — Across five separate testing days, subjects were administered two placebo doses, 20 mg damphetamine,150 mg caffeine, and 300 mg caffeine in counterbalanced fashion
  Other Names: Vivarin
  Arms: 4 Caffeine 300 mg

SUMMARY:
This study is being done to find out if medicines that affect a neurotransmitter (chemical messenger) in the brain called adenosine improve behavioral problems that are related to drug abuse. Another purpose of the study is to find out how genes related to adenosine change how people respond to these medicines. More information about how these medicines change behaviors may be helpful to come up with new treatments for drug abuse.

DETAILED DESCRIPTION:
Specific Aims:

Aim 1. To characterize the behavioral and subjective effects of acute caffeine administration in cocaine-dependent subjects, using laboratory measures of impulse control, drug discrimination (with d-amphetamine as the training dose), and subjective effects.

Hypotheses related to Aim 1:

1. Subjects will show decreases in impulsivity (delay to reward and response inhibition) after acute oral doses of caffeine compared to placebo.
2. Subjects will show some stimulant-like subjective effects following acute oral doses of caffeine, but not the euphoric effects that would predict abuse potential.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who currently meet DSM-IV criteria for cocaine dependence and healthy controls
* At least one cocaine positive urine during screening.
* Current regular consumption of caffeine.
* Female subjects: a negative pregnancy test.

Exclusion Criteria:

* Current or past DSM-IV Axis I disorder other than substance abuse/ dependence
* Any significant non-psychiatric medical illness requiring ongoing medical treatment or which would preclude treatment with d-amphetamine or caffeine
* Substance dependence other than cocaine within the last 3 months.
* Positive breath alcohol.
* Positive urine drug screen for drugs other than cocaine or THC at the time of behavioral testing
* For female subjects: known pregnancy or a positive pregnancy test or current breast feeding.
* Diagnosis of Adult Attention Deficit Disorder as determined by: a) meeting DSM-IV criteria for childhood ADHD, b) currently has impairing ADHD symptoms, c) ADHD symptoms can not have remitted at any period since childhood.
* HIV positive.
* I.Q. below 70.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2008-04; Primary Completion 2011-07 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick G Moeller, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center, Houston, Houston, Texas, United States

REFERENCES:
- [Result] Lane SD, Green CE, Schmitz JM, Rathnayaka N, Fang WB, Ferre S, Moeller FG. Comparison of Caffeine and d-amphetamine in Cocaine-Dependent Subjects: Differential Outcomes on Subjective and Cardiovascular Effects, Reward Learning, and Salivary Paraxanthine. J Addict Res Ther. 2014;5(2):176. doi: 10.4172/2155-6105.1000176. PMID 25414797

RESULTS

PARTICIPANT FLOW:
Groups:
- Cocaine Users: Cocaine users were allocated to different sequence orders for the 5 interventions
  Across five separate testing days, subjects were administered two placebo doses, 20 mg amphetamine, 150 mg caffeine, and 300 mg caffeine in counterbalanced fashion
- Control Participants: Control participants were allocated to different sequence orders for the 5 interventions
  Across five separate testing days, subjects were administered two placebo doses, 20 mg amphetamine, 150 mg caffeine, and 300 mg caffeine in counterbalanced fashion
Period: Overall Study
Arm/Group | Cocaine Users | Control Participants
Started | 13 | 10
Completed | 13 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cocaine Users: Across five separate testing days, subjects were administered two placebo doses, 20 mg amphetamine, 150 mg caffeine, and 300 mg caffeine in counterbalanced fashion
- Control Participants: Across five separate testing days, subjects were administered two placebo doses, 20 mg amphetamine,150 mg caffeine, and 300 mg caffeine in counterbalanced fashion
- Total: Total of all reporting groups
Arm/Group | Cocaine Users | Control Participants | Total
Number analyzed (Participants) | 13 | 10 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 10 | 23
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 10 | 5 | 15
Region of Enrollment [Number; unit: participants]
  United States | 13 | 10 | 23

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale Subjective Rating of Drug Effects
Description: Visual Analog Scale Rating. Scores range from 0 to 100 with higher scores meaning greater intensity of response being rated.
Time Frame: Immediately after dose
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: Placebo
  Placebo: Across five separate testing days, subjects were administered two placebo doses, 20 mg amphetamine, 150 mg caffeine, and 300 mg caffeine in counterbalanced fashion
- Caffeine 150 Mg: 150 MG of Caffeine
- Caffeine 300 mg: Caffeine 300 mg
- Amphetamine 20 mg: Amphetamine 20 mg
Arm/Group | Placebo | Caffeine 150 Mg | Caffeine 300 mg | Amphetamine 20 mg
Number analyzed (Participants) | 23 | 23 | 23 | 23
units on a scale
  Elation: Control (N=10) | 8.65 (5.33) | 9.85 (5.32) | 13.65 (6.1) | 10.43 (4.48)
  Elation: Cocaine (N=13) | 25.99 (6.01) | 32.54 (7.62) | 21.65 (5.68) | 25.71 (6.42)
  Anxious: Control (N=10) | 10.15 (5.31) | 10.45 (5.69) | 8.50 (4.91) | 11.68 (4.62)
  Anxious: Cocaine (N=13) | 19.64 (6.17) | 21.35 (6.01) | 25.27 (7.12) | 21.71 (5.43)
  Vigor: Control (N=10) | 8.25 (2.06) | 8.50 (1.92) | 9.78 (1.98) | 8.28 (2.01)
  Vigor: Cocaine (N=13) | 10.42 (1.54) | 10.85 (1.59) | 9.27 (1.60) | 10.31 (1.33)
  Tension: Control (N=10) | 1.05 (0.38) | 1.60 (0.53) | 1.62 (0.60) | 1.53 (0.48)
  Tension: Cocaine (N=13) | 1.63 (0.62) | 0.96 (0.57) | 2.38 (0.94) | 1.88 (0.61)
  Fatigue: Control (N=10) | 3.85 (1.37) | 3.00 (1.48) | 3.44 (1.64) | 3.60 (1.07)
  Fatigue: Cocaine (N=13) | 0.68 (0.32) | 0.54 (0.25) | 1.69 (0.71) | 1.17 (0.36)
  Depression: Control (N=10) | 0.10 (0.10) | 0.10 (0.10) | 0.41 (0.30) | 0.10 (0.06)
  Depression: Cocaine (N=13) | 1.05 (0.54) | 0.62 (0.47) | 1.96 (1.12) | 1.10 (0.51)

2. Primary Outcome: Systolic and Diastolic Blood Pressure
Description: Sitting Blood Pressure
Time Frame: Average across 7 time points: Immediately after dose and every 30 minutes for 3 hours
Measure: Mean (Standard Error); unit: mmHg
Groups:
- Caffeine 300 mg: Caffeine 300mg
- Amphetamine 20mg: Amphetamine 20mg
Arm/Group | Placebo | Caffeine 150 Mg | Caffeine 300 mg | Amphetamine 20mg
Number analyzed (Participants) | 23 | 23 | 23 | 23
mmHg
  SBP Control (N=10) | 115.64 (3.41) | 115.9 (4.07) | 117.36 (4.2) | 119.27 (2.13)
  SBP Cocaine (N=13) | 120.18 (1.40) | 122.10 (1.81) | 123.84 (2.18) | 120.30 (1.58)
  DBP Control (N=10) | 74.82 (2.78) | 75.33 (2.72) | 77.94 (1.42) | 77.83 (1.45)
  DBP Cocaine (N=13) | 79.66 (3.01) | 79.98 (1.79) | 82.81 (1.74) | 78.16 (1.56)

3. Primary Outcome: Heart Rate
Description: Sitting heart rate
Time Frame: Average across 7 time points: Immediately after dose and every 30 minutes for 3 hours
Measure: Mean (Standard Error); unit: Beats per minute
Arm/Group | Placebo | Caffeine 150 Mg | Caffeine 300 mg | Amphetamine 20mg
Number analyzed (Participants) | 23 | 23 | 23 | 23
Beats per minute
  Control (N=10) | 66.10 (1.88) | 62.47 (2.09) | 61.33 (1.67) | 65.55 (1.23)
  Cocaine (N=13) | 63.08 (2.11) | 62.60 (3.00) | 61.57 (1.40) | 63.51 (2.99)

4. Primary Outcome: Addiction Research Center Inventory Subjective Rating of Drug Effects
Description: Addiction Research Center Inventory (ARCI 49). T/F scales with 49 items.
  Includes the following subscales:
  Morphine-Benzedrine Group (MBG), includes euphoria (0 to +16, higher numbers = more euphoria) Phenobarbital-Chorpromazine-Alcohol Group (PCAG), includes sedation (-3 to +11, higher scores = more sedation) Lysergic Acid Diethylmide Group (LSD) , includes dysphoria and agitation (-4 to +10, higher scores = more dysphoria) Amphetamine Group (A), includes stimulation ( 0 to +11, higher scores = more stimulation) Benzedrine Group (BG), includes energy and "intellectual efficiacy" (+4 to +9, higher scores = more energy)
Time Frame: Immediately after dose
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Caffeine 150 Mg | Caffeine 300 mg | Amphetamine 20 mg
Number analyzed (Participants) | 23 | 23 | 23 | 23
units on a scale
  PCAG: Control (N=10) | 3.87 (0.82) | 3.62 (0.83) | 3.52 (0.79) | 3.64 (0.71)
  PCAG: Cocaine (N=13) | 1.95 (0.58) | 1.83 (0.68) | 2.95 (0.82) | 2.43 (0.67)
  A: Control (N=10) | 3.20 (0.51) | 3.60 (0.68) | 3.80 (0.59) | 3.22 (0.38)
  A: Cocaine (N=13) | 3.30 (0.51) | 3.39 (0.54) | 3.19 (0.44) | 3.69 (0.45)
  BG: Control (N=10) | 6.00 (0.39) | 6.35 (0.56) | 6.05 (0.57) | 5.83 (0.36)
  BG: Cocaine (N=13) | 5.69 (0.34) | 5.77 (0.37) | 5.07 (0.61) | 5.57 (0.51)
  MGB: Control (N=10) | 4.09 (1.26) | 4.34 (1.31) | 5.14 (1.37) | 4.04 (1.28)
  MGB: Cocaine (N=13) | 5.29 (1.13) | 5.62 (1.23) | 4.31 (0.96) | 5.18 (1.00)
  LSD: Control (N=10) | 1.78 (0.44) | 2.43 (0.56) | 1.23 (0.41) | 1.70 (0.41)
  LSD: Cocaine (N=13) | 0.89 (0.47) | 0.48 (0.49) | 1.05 (0.49) | 0.98 (0.45)

5. Primary Outcome: Drug Effects Questionnaire Rating of Subjective Ratings of Drug Effects
Description: Assessments measured using a 4 item Drug Effects Questionnaire (DEQ) Ranges from 0 to 100 with higher numbers showing greater effect for each scale.
Time Frame: Immediately after dose
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Caffeine 150 Mg | Caffeine 300 mg | Amphetamine 20 mg
Number analyzed (Participants) | 23 | 23 | 23 | 23
units on a scale
  Feel effects:Control (N=10) | 16.75 (7.58) | 20.25 (6.31) | 9.45 (4.97) | 11.37 (4.93)
  Feel effects:Cocaine (N=13) | 17.30 (5.80) | 20.73 (5.95) | 17.62 (5.91) | 18.68 (6.08)
  Like effects:Control (N=10) | 39.92 (6.82) | 35.62 (6.89) | 52.17 (6.95) | 42.25 (5.74)
  Like effects:Cocaine (N=13) | 37.18 (9.74) | 39.94 (10.55) | 43.75 (7.21) | 32.04 (8.63)
  High:Control (N=10) | 10.77 (5.23) | 12.17 (5.59) | 7.17 (4.16) | 7.17 (3.95)
  High:Cocaine (N=13) | 14.35 (5.45) | 16.14 (5.67) | 15.87 (5.78) | 14.64 (5.44)
  Like more:Control (N=10) | 25.77 (7.20) | 25.62 (6.54) | 32.92 (7.01) | 25.65 (6.08)
  Like more:Cocaine (N=13) | 25.96 (9.18) | 25.68 (8.99) | 28.71 (8.48) | 26.16 (8.69)

6. Secondary Outcome: Probabalistic Feedback Selection Task
Description: Accuracy on a range from 0 to 1 of correctly performing a learning task, with 1 being the highest degree of accuracy.
Time Frame: 75 minutes after dose
Measure: Mean (Standard Error); unit: accuracy
Arm/Group | Placebo | Caffeine 150 Mg | Caffeine 300 mg | Amphetamine 20mg
Number analyzed (Participants) | 23 | 23 | 23 | 23
accuracy
  Control (N=10) | 0.56 (0.02) | 0.55 (0.03) | 0.56 (0.02) | 0.61 (0.02)
  Cocaine (N=13) | 0.54 (0.01) | 0.56 (0.02) | 0.58 (0.02) | 0.56 (0.02)

7. Secondary Outcome: Saliva Caffeine and Paraxanthine Levels
Description: Due to insufficient oral volume or breakage during sample transfer, data were lost or incomplete for two cocaine-dependent subjects.
  Analyses for the saliva data represent 11 cocaine-dependent subjects and 10 controls.
Time Frame: 30 minutes prior to dose, 30/90/150 minutes post dose.
Population: Assessment was not performed for amphetamine intervention
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo | Caffeine 150 Mg | Caffeine 300 mg | Amphetamine 20mg
Number analyzed (Participants) | 21 | 21 | 21 | 0
ng/mL
  Caffeine -30 min Control (N=10) | 1000 (490) | 510 (470) | 335 (110) |
  Caffeine 30 min Control (N=10) | 983 (440) | 2715 (1110) | 2895 (998) |
  Caffeine 90 min Control (N=10) | 984 (445) | 2225 (995) | 3510 (1001) |
  Caffeine 150 min Control (N=10) | 984 (601) | 1910 (898) | 3270 (901) |
  Caffeine -30 min Cocaine (N=11) | 990 (920) | 998 (820) | 1201 (997) |
  Caffeine 30 min Cocaine (N=11) | 780 (510) | 2125 (1001) | 3510 (1220) |
  Caffeine 90 min Cocaine (N=11) | 625 (410) | 2077 (874) | 3720 (911) |
  Caffeine 150 min Cocaine (N=11) | 510 (322) | 1909 (605) | 3205 (697) |
  Parathanxine -30 min Control (N=10) | 440 (155) | 274 (140) | 198 (92) |
  Parathanxine 30 min Control (N=10) | 410 (240) | 301 (238) | 202 (101) |
  Parathanxine 90 min Control (N=10) | 411 (219) | 402 (155) | 397 (110) |
  Parathanxine 150 min Control (N=10) | 410 (143) | 411 (145) | 462 (215) |
  Parathanxine -30 min Cocaine (N=11) | 334 (205) | 401 (197) | 408 (240) |
  Parathanxine 30 min Cocaine (N=11) | 320 (275) | 465 (185) | 656 (280) |
  Parathanxine 90 min Cocaine (N=11) | 321 (248) | 601 (233) | 985 (245) |
  Parathanxine 150 min Cocaine (N=11) | 296 (252) | 605 (247) | 1014 (255) |

ADVERSE EVENTS:
Groups:
- 1 Caffeine: Caffeine
  Caffeine: Across five separate testing days, subjects were administered two placebo doses, 20 mg amphetamine, 150 mg caffeine, and 300 mg caffeine in counterbalanced fashion
Arm/Group | 1 Caffeine | 2 Placebo | 3 Amphetamine
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No